CLINICAL TRIAL: NCT02806947
Title: A Randomized, Phase II, Multicenter, Open Label, Study Evaluating Sirolimus and Prednisone in Patients With Refined Minnesota Standard Risk, Ann Arbor 1/2 Confirmed Acute Graft-Versus-Host Disease (BMT CTN 1501)
Brief Title: A Study to Evaluate Steroid-free Treatment for Standard-Risk aGVHD (BMT CTN 1501)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMT CTN 1501; 2U10HL069294-11 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2016-06-08; First posted 2016-06-21 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2019-06

CONDITIONS: Acute GVHD
Keywords: Acute GVHD; Standard-Risk; Sirolimus; Refined Minnesota Risk Criteria; Ann Arbor; Biomarker; Steroid-Free
MeSH Terms: interventions — Sirolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus (Experimental): Sirolimus, a steroid-free therapy, will be administered after a diagnosis of standard-risk aGVHD is clinically established.
  Interventions: Drug: Sirolimus
- Prednisone (Active Comparator): Prednisone, standard of care therapy for GVHD, will be administered after a diagnosis of standard-risk aGVHD is clinically established.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Sirolimus — Sirolimus will be administered with a starting dose of 6 mg for patients older than 12 years, or 5 mg/m^2 for patients ≤ 12 years. Trough levels will be routinely measured and sirolimus will be kept at maintenance dosing for target therapeutic levels for minimum duration through Day 56 post-randomization.
  Other Names: Rapamycin; Rapamune®
  Arms: Sirolimus
Drug: Prednisone — Prednisone will be administered at 2mg/kg/day x 3 days, and then tapered according to individual treating clinician judgment.
  Other Names: Deltasone®; Orasone®; Cortan®; Sterapred®
  Arms: Prednisone

SUMMARY:
The study is a Phase II randomized, open label, multicenter trial designed to identify whether sirolimus is a potential alternative to prednisone as an up-front treatment for patients with standard-risk acute GVHD defined according to clinical and biomarker-based risk stratification. This trial incorporates both a novel up front GVHD therapy (sirolimus) as well as a novel BMT CTN developed acute GVHD biomarker test.

DETAILED DESCRIPTION:
The study is a Phase II randomized, open label, multicenter trial designed to identify whether sirolimus is a potential alternative to prednisone as an up-front treatment for patients with standard-risk acute GVHD defined according to clinical and biomarker-based risk stratification.

Patients with previously untreated, standard-risk acute GVHD, according to the refined Minnesota Criteria, who are in need of systemic therapy, will have a 5 mL blood sample collected prior to randomization to assess their biomarker Ann Arbor Risk status. Ann Arbor scoring results will be provided 48-72 hours after randomization. Patients will begin their study treatment assignments within 24 hours of randomization. Those with biomarker results of combined AA1/2 risk will continue on their randomized study treatment and will be included for primary endpoint analysis (Day 28 complete or partial response) and all planned study procedures and assessments. In contrast, patients with AA3 biomarker risk and those patients with missing biomarker results may continue on their randomized therapies or start another therapy at their physicians' discretion. In addition, AA3 risk patients and those with missing results will not be considered in primary endpoint analysis, but will be included in a subset analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with standard-risk acute GVHD, according to refined Minnesota Criteria. Refined Minnesota Criteria are available at https://redcap.ahc.umn.edu/surveys/?s=bNmFhseJIf.

   Standard-risk acute GVHD according to the refined Minnesota Risk Criteria requires meeting one of the criteria below:
   1. Single organ involvement (Stage 1-3 skin, Stage 1 upper GI, or Stage 1-2 lower GI)
   2. Multiple organ involvement (Stage 1-3 skin plus stage 1 upper GI, Stage 1-3 skin plus stage 1 lower GI, Stage 1-3 skin plus stage 1 lower GI plus stage 1 upper GI, Stage 1-3 skin plus stage 1-4 liver, or Stage 1 lower GI plus stage 1 upper GI)
2. Acute Minnesota Standard Risk GVHD requiring systemic immune suppressive therapy.
3. Acute GVHD developing after allogeneic hematopoietic cell transplantation using either bone marrow, peripheral blood, or umbilical cord blood. Recipients of non-myeloablative, reduced intensity conditioning and myeloablative transplants are eligible. All allogeneic donor sources are permitted, including siblings, unrelated donors, human leukocyte antigen (HLA)-haploidentical related donors and umbilical cord blood.
4. Patients NOT receiving systemic immune suppressive therapy for treatment of active GVHD (topical skin and GI corticosteroids are allowed).
5. Ability to tolerate oral or enterically-administered medications.
6. Patients of all ages.
7. Absolute neutrophil count (ANC) greater than 500/µL.
8. Biopsy confirmation of GVHD is not required. Enrollment should not be delayed for biopsy or pathology results unless local institutional practice mandates biopsy confirmation to make a GVHD treatment decision.
9. Written informed consent and/or assent from patient, parent or guardian.
10. Collection of a 5 ml blood sample (red top for serum) from the patient for Ann Arbor Scoring and ready to be shipped immediately after randomization.

Exclusion Criteria:

1. Patients receiving sirolimus (for any indication including GVHD prophylaxis) within 14 days of screening for enrollment.
2. Relapsed, progressing or persistent malignancy requiring withdrawal of systemic immune suppression.
3. Patients with acute GVHD developing after a donor lymphocyte infusion.
4. Active or recent (within 7 days) episode of transplant associated microangiopathy.
5. Patients with uncontrolled infections will be excluded. Infections are considered controlled if appropriate therapy has been instituted and, at the time of enrollment, no signs of progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
6. Patients unlikely to be available for evaluation at the transplant center on Day 28 and 56 of therapy.
7. A clinical presentation resembling de novo chronic GVHD or overlap syndrome developing before or present at the time of enrollment.
8. Patients receiving corticosteroids for any indication within 7 days before the onset of acute GVHD, except the following: Stable replacement doses of corticosteroids for adrenal insufficiency are permitted (e.g. hydrocortisone total dose of 10-12 mg/m^2/day or prednisone 5-7.5mg daily or equivalent). Corticosteroids administered as premedication before transfusion of blood products or before intravenous medications to prevent infusion reactions are allowed.
9. Patients who are pregnant or breastfeeding.
10. Females of childbearing potential (FCBP) or a man who has sexual contact with a FCBP and is unwilling to use effective birth control for the duration of the study.
11. Patients on dialysis.
12. Patients on mechanical ventilation.
13. Patients with severe hepatic sinusoidal obstruction syndrome who in the judgment of the treating physician are not expected to have normalized bilirubin by Day 56 after enrollment.
14. Patients with a history of hypersensitivity to sirolimus or any component of the formulation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research
Locations (21):
- United States (21):
  - City of Hope National Medical Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Blood & Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas/MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University MCV Hospitals, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Derived] Giaccone L, Faraci DG, Butera S, Lia G, Di Vito C, Gabrielli G, Cerrano M, Mariotti J, Dellacasa C, Felicetti F, Brignardello E, Mavilio D, Bruno B. Biomarkers for acute and chronic graft versus host disease: state of the art. Expert Rev Hematol. 2021 Jan;14(1):79-96. doi: 10.1080/17474086.2021.1860001. Epub 2020 Dec 24. PMID 33297779
- [Derived] Pidala J, Hamadani M, Dawson P, Martens M, Alousi AM, Jagasia M, Efebera YA, Chhabra S, Pusic I, Holtan SG, Ferrara JLM, Levine JE, Mielcarek M, Anasetti C, Antin JH, Bolanos-Meade J, Howard A, Logan BR, Leifer ES, Pritchard TS, Horowitz MM, MacMillan ML. Randomized multicenter trial of sirolimus vs prednisone as initial therapy for standard-risk acute GVHD: the BMT CTN 1501 trial. Blood. 2020 Jan 9;135(2):97-107. doi: 10.1182/blood.2019003125. PMID 31738834

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The primary analysis population includes only participants with an AA score of 1 or 2 (n=64 on the prednisone arm, n=58 on the sirolimus arm). Three participants on the prednisone arm and two on the sirolimus arm were excluded because they had an AA score of 3 or missing.
Period: Overall Study
Arm/Group | Sirolimus | Prednisone
Started | 58 | 64
Completed | 53 | 63
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus | Prednisone | Total
Number analyzed (Participants) | 58 | 64 | 122
Age, Continuous [Median (Full Range); unit: years] | 58.0 [7.8 to 74.7] | 52.4 [0.9 to 72.7] | 54.6 [0.9 to 74.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 31 | 52
  Male | 37 | 33 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian / Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Hawaiian/Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 55 | 59 | 114
  Multiracial | 0 | 0 | 0
  Unknown | 1 | 2 | 3
Ann Arbor Biomarker Risk Score [Count of Participants; unit: Participants] — The Ann Arbor biomarker risk score is a scoring system for predicting risk of non-relapse mortality in patients with graft versus host disease. Risk is classified as 1, 2, or 3, where 1 denotes the lowest risk and 3 the highest risk.
  Participants
    1 | 38 | 45 | 83
    2 | 20 | 19 | 39
Skin Abnormalities at Enrollment [Count of Participants; unit: Participants] — Abnormalities in skin that are characteristics of graft versus host disease (GVHD) are tabulated.
  Participants
    No active GVHD rash | 20 | 19 | 39
    Maculopapular Rash <25% body surface area | 8 | 11 | 19
    Maculopapular Rash 25-50% body surface area | 14 | 13 | 27
    Maculopapular Rash >50% body surface area | 16 | 21 | 37
Upper GI Abnormalities at Enrollment [Count of Participants; unit: Participants] — Abnormalities in the upper GI tract that are characteristics of graft versus host disease (GVHD) are tabulated.
  Participants
    No or Intermittent Nausea, Vomiting, or Anorexia | 32 | 36 | 68
    Persistent Nausea, Vomiting, or Anorexia | 26 | 28 | 54
Lower GI Abnormalities at Enrollment [Count of Participants; unit: Participants] — Diarrhea volume is tabulated, as diarrhea is characteristics of graft versus host disease (GVHD).
  Participants
    No Diarrhea | 53 | 46 | 99
    Adult: <500 mL/day, Child: <10mL/kg/day | 3 | 10 | 13
    Adult: 500-999mL/day, Child: 10-19.9mL/kg/day | 2 | 7 | 9
    Adult: 1000-1500mL/day, Child: 20-30mL/kg/day | 0 | 1 | 1
Liver Abnormalities at Enrollment [Count of Participants; unit: Participants] — Abnormalities in the liver that are characteristics of graft versus host disease (GVHD) are tabulated.
  Participants
    Bilirubin <2.0mg/dL | 58 | 63 | 121
    Bilirubin 2.0-3.0mg/dL | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete or Partial Response (CR/PR) to Acute GVHD Treatment
Description: Scoring of CR/PR is in comparison to the participant's acute GVHD status at randomization. Complete response (CR) is defined as staging of 0 for in all target organs for GVHD - skin, GI tract, and liver. Partial response (PR) is defined as improvement in some target organ(s) without worsening in others. Death and initiation of systemic acute GVHD treatment beyond randomized treatment are considered failures for this endpoint. Organ staging is defined below:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area (BSA)
  2. Rash on 25-50% of BSA
  3. Rash on >50% of BSA
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level):
  0: <2 mg/dL
  1. 2-3 mg/dL
  2. 3.01-6 mg/dL
  3. 6.01-15.0 mg/dL
  4. >15 mg/dL
  GI stage:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus
Time Frame: Days 28 and 56 Post-randomization
Population: CR/PR was evaluated in participants remaining on study until the assessment time point. At Day 28, one prednisone and four sirolimus arm participants were excluded from the analysis due to prior study withdrawal. At Day 56, one prednisone and five sirolimus arm participants were excluded from the analysis due to prior study withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
Participants
  CR/PR at Day 28: number analyzed (Participants) | 54 | 63
  CR/PR at Day 28: Yes | 35 | 46
  CR/PR at Day 28: No | 19 | 17
  CR/PR at Day 56: number analyzed (Participants) | 53 | 63
  CR/PR at Day 56: Yes | 34 | 50
  CR/PR at Day 56: No | 19 | 13
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The primary objective of this Phase II trial was to describe the proportion of patients with Day 28 CR/PR in each treatment arm and to estimate the risk difference of these rates using a point estimate and 90% confidence interval. These estimates are used to inform about the efficacy of sirolimus in contrast to prednisone for potential future research; Test type: Other — No formal hypothesis test was planned or performed for comparing Day 28 CR/PR proportions between arms. Rather, the risk difference is estimated by a point estimate and 90% confidence interval; Risk Difference (RD) = -0.082, 90% CI 2-sided [-0.223 to 0.059], Standard Error of Mean 0.086 — The risk difference estimate is the observed proportion of Day 28 CR/PR in the sirolimus arm minus the proportion in the prednisone arm. A Wald confidence interval for this difference is given
Statistical Analysis 2: Comparison: Sirolimus vs Prednisone; A secondary objective of this Phase II trial was to describe the proportion of patients with Day 56 CR/PR in each treatment arm and to estimate the risk difference of these rates using a point estimate and 95% confidence interval. These estimates are used to inform about the efficacy of sirolimus in contrast to prednisone for potential future research; Test type: Other — No formal hypothesis test was planned or performed for comparing Day 56 CR/PR proportions between arms. Rather, the risk difference is estimated by a point estimate and 95% confidence interval; Risk Difference (RD) = -0.152, 95% CI 2-sided [-0.315 to 0.011], Standard Error of Mean 0.083 — The risk difference estimate is the observed proportion of Day 56 CR/PR in the sirolimus arm minus the proportion in the prednisone arm. A Wald confidence interval for this difference is given

2. Secondary Outcome: Percentage of Participants With Complete or Partial Response (CR/PR) and Steroid Dose Less Than 0.25 mg/kg Per Day
Description: The proportion of patients with CR/PR and on a prednisone-equivalent steroid dose of 0.25 mg/kg/day or less is evaluated. CR/PR scoring is in comparison to acute GVHD status at randomization. CR is defined as staging of 0 in all target organs. PR is defined as improvement in some organ(s) without worsening in others. Death and initiation of steroid-free, systemic acute GVHD treatment beyond randomized therapy are considered failures for this endpoint. Organ staging is defined as:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area (BSA)
  2. Rash 25-50% of BSA
  3. Rash >50% of BSA
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level in mg/dL):
  0: <2
  1. 2-3
  2. 3.01-6
  3. 6.01-15.0
  4. >15 mg/dL
  GI stage:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus
Time Frame: Day 28 Post-randomization
Population: The endpoint was evaluated only in participants that remained on study until Day 28. One participant on the prednisone arm and four on the sirolimus arm were deemed unevaluable at Day 28 due to prior study withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 54 | 63
Participants
  Yes | 36 | 20
  No | 18 | 43
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with CR/PR and steroid dose of 0.25mg/kg/day or less at Day 28 post-randomization between the sirolimus and prednisone arms. These proportions were compared between treatment arms using a Z test of the difference of binomial proportions; Test type: Superiority; p < 0.001, Z test comparing binomial proportions — Statistical significance was determined using a pre-specified threshold of 0.05

3. Secondary Outcome: Acute GVHD Response
Description: Acute GVHD response is classified as CR, PR, mixed response (MR), no response (NR), and progression and scored by comparison to acute GVHD status at randomization. MR is defined as improvement in some organ(s) with worsening in another, progression as worsening in some organ(s) without improvement in others, and NR as absence of any improvement or worsening. Death and initiation of systemic acute GVHD treatment beyond randomized treatment are classified as NR. Organ staging is defined as:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area (BSA)
  2. Rash 25-50% of BSA
  3. Rash >50% of BSA
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level in mg/dL):
  0: <2
  1. 2-3
  2. 3.01-6
  3. 6.01-15.0
  4. >15
  GI stage:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus
Time Frame: Days 28 and 56 Post-randomization
Population: Acute GVHD response was evaluated in participants remaining on study until the assessment day. At Day 28, one prednisone and four sirolimus arm participants were excluded from the analysis due to prior study withdrawal. At Day 56, one prednisone and five sirolimus arm participants were excluded from the analysis due to prior study withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
Participants
  Acute GVHD Response at Day 28: number analyzed (Participants) | 54 | 63
  Acute GVHD Response at Day 28: Complete Response (CR) | 30 | 39
  Acute GVHD Response at Day 28: Partial Response (PR) | 5 | 7
  Acute GVHD Response at Day 28: Mixed Response (MR) | 1 | 5
  Acute GVHD Response at Day 28: No Response (NR) | 16 | 11
  Acute GVHD Response at Day 28: Progression | 2 | 1
  Acute GVHD Response at Day 56: number analyzed (Participants) | 53 | 63
  Acute GVHD Response at Day 56: Complete Response (CR) | 30 | 48
  Acute GVHD Response at Day 56: Partial Response (PR) | 4 | 2
  Acute GVHD Response at Day 56: Mixed Response (MR) | 0 | 0
  Acute GVHD Response at Day 56: No Response (NR) | 19 | 10
  Acute GVHD Response at Day 56: Progression | 0 | 3
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in classification of acute GVHD response at Day 28 post-randomization between participants on the sirolimus and prednisone arms. These classifications were compared between treatment arms using Fisher's exact test, due to the presence of small numbers of participants in some categories; Test type: Superiority; p = 0.320, Fisher Exact — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in classification of acute GVHD response at Day 56 post-randomization between participants on the sirolimus and prednisone arms. These classifications were compared between treatment arms using Fisher's exact test, due to the presence of small numbers of participants in some categories; Test type: Superiority; p = 0.014, Fisher Exact — Statistical significance was determined using a pre-specified threshold of 0.05

4. Secondary Outcome: Percentage of Participants With Treatment Failure
Description: Treatment failure is defined as either no response (NR) or progression and scored by comparison to acute GVHD status at randomization. Progression is defined as worsening in some target organ(s) without improvement in others and NR is defined as absence of any improvement or worsening in target organs. Death and initiation of systemic acute GVHD treatment beyond randomized treatment are classified as NR. Organ staging is defined as:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area (BSA)
  2. Rash 25-50% of BSA
  3. Rash >50% of BSA
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level in mg/dL):
  0: <2
  1. 2-3
  2. 3.01-6
  3. 6.01-15.0
  4. >15
  GI stage:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus
Time Frame: Days 28 and 56 Post-randomization
Population: Treatment failure was evaluated in participants remaining on study until the assessment day. At Day 28, one prednisone and four sirolimus arm participants were excluded from the analysis due to prior study withdrawal. At Day 56, one prednisone and five sirolimus arm participants were excluded from the analysis due to prior study withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
Participants
  Treatment Failure at Day 28: number analyzed (Participants) | 54 | 63
  Treatment Failure at Day 28: Yes | 18 | 12
  Treatment Failure at Day 28: No | 36 | 51
  Treatment Failure at Day 56: number analyzed (Participants) | 53 | 63
  Treatment Failure at Day 56: Yes | 19 | 13
  Treatment Failure at Day 56: No | 34 | 50
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with treatment failure at Day 28 post-randomization between the sirolimus and prednisone arms. These proportions were compared between treatment arms using a Z test of the difference of binomial proportions; Test type: Superiority; p = 0.078, Z test comparing binomial proportions — Statistical significance was determine using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with treatment failure at Day 56 post-randomization between the sirolimus and prednisone arms. These proportions were compared between treatment arms using a Z test of the difference of binomial proportions; Test type: Superiority; p = 0.068, Z test comparing binomial proportions — Statistical significance was determined using a pre-specified threshold of 0.05

5. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Overall survival is defined as survival of death from any cause.
Time Frame: 6 and 12 Months Post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
percentage of participants
  Overall Survival at 6 Months | 81.9 [68.9 to 89.8] | 82.7 [71.0 to 90.0]
  Overall Survival at 12 Months | 76.3 [62.7 to 85.5] | 73.2 [60.4 to 82.4]
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with overall survival between the sirolimus and prednisone arms during the 12 month period post-randomization. These proportions were compared between treatment arms using a log rank test; Test type: Superiority; p = 0.785, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05

6. Secondary Outcome: Percentage of Participants With Disease-free Survival
Description: Disease-free survival is defined as freedom from death and relapse of the underlying malignancy.
Time Frame: 6 and 12 Months Post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
percentage of participants
  Disease-free Survival at 6 Months | 72.8 [58.9 to 82.6] | 78.1 [65.9 to 86.4]
  Disease-free Survival at 12 Months | 61.6 [47.4 to 73.0] | 70.2 [57.3 to 79.8]
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with disease-free survival between the sirolimus and prednisone arms during the 12 month period post-randomization. These proportions were compared between treatment arms using a log rank test; Test type: Superiority; p = 0.340, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05

7. Secondary Outcome: Proportion of Participants With Event-free Survival
Description: Event-free survival is defined as freedom from acute GVHD progression, chronic GVHD, malignancy relapse, and death.
Time Frame: 6 and 12 Months Post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
percentage of participants
  Event-free Survival at 6 Months | 47.3 [33.6 to 59.7] | 43.7 [31.4 to 55.4]
  Event-free Survival at 12 Months | 35.9 [23.4 to 48.5] | 31.2 [20.4 to 42.7]
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with event-free survival between the sirolimus and prednisone arms during the 12 month period post-randomization. These proportions were compared between treatment arms using a log rank test; Test type: Superiority; p = 0.713, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05

8. Secondary Outcome: Percentage of Participants With Non-relapse Mortality
Description: Non-relapse mortality is defined as death due to any cause other than relapse of the underlying malignancy. The cumulative incidence of non-relapse mortality is described, with malignancy relapse treated as a competing risk.
Time Frame: 6 and 12 Months Post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
percentage of participants
  Non-relapse Mortality at 6 Months | 12.7 [5.5 to 23.0] | 9.4 [3.8 to 18.1]
  Non-relapse Mortality at 12 Months | 16.5 [8.1 to 27.6] | 14.2 [6.9 to 24.0]
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with non-relapse mortality between the sirolimus and prednisone arms during the 12 month period post-randomization, with malignancy relapse treated as a competing risk for non-relapse mortality. These proportions were compared between treatment arms using Gray's test; Test type: Superiority; p = 0.726, Gray's test — Statistical significance was determined using a pre-specified threshold of 0.05

9. Secondary Outcome: Percentage of Participants With Malignancy Relapse
Description: The cumulative incidence of relapse of the primary malignancy is described, with death treated as a competing risk.
Time Frame: 6 and 12 Months Post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
percentage of participants
  Malignancy Relapse at 6 Months | 14.5 [6.7 to 25.1] | 12.5 [5.8 to 21.9]
  Malignancy Relapse at 12 Months | 21.9 [12.0 to 33.7] | 15.7 [8.0 to 25.7]
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with malignancy relapse between the sirolimus and prednisone arms during the 12 month period post-randomization, with death treated as a competing risk for malignancy relapse. These proportions were compared between treatment arms using Gray's test; Test type: Superiority; p = 0.402, Gray's test — Statistical significance was determined using a pre-specified threshold of 0.05

10. Secondary Outcome: Percentage of Participants With Chronic GVHD
Description: Chronic GVHD is classified per 2005 NIH Consensus Criteria (Filipovich et al. 2005) into categories of severity: none, mild, moderate, and severe. Occurrence of chronic GVHD is defined as the occurrence of mild, moderate, or severe chronic GVHD per this classification. The cumulative incidence of chronic GVHD is described, with death and malignancy relapse treated as competing risks.
Time Frame: 6 and 12 Months Post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
percentage of participants
  Chronic GVHD at 6 Months | 25.7 [14.9 to 37.9] | 31.2 [20.2 to 42.8]
  Chronic GVHD at 12 Months | 31.4 [19.5 to 44.0] | 40.6 [28.4 to 52.4]
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with chronic GVHD between the sirolimus and prednisone arms during the 12 month period post-randomization, with death and malignancy relapse treated as competing risks for chronic GVHD. These proportions were compared between treatment arms using Gray's test; Test type: Superiority; p = 0.296, Gray's test — Statistical significance was determined using a pre-specified threshold of 0.05

11. Secondary Outcome: Percentage of Participants With GVHD-free Survival
Description: GVHD-free survival is defined as freedom from acute GVHD, chronic GVHD, and death. The proportion of participants alive and free of both acute and chronic GVHD are described at 6 and 12 months post-randomization.
Time Frame: 6 and 12 Months Post-randomization
Population: GVHD-free survival was evaluated only in participants that remained on study until the assessment time point. One participant on the prednisone arm and five on the sirolimus arm were excluded from the analysis at 6 and 12 months due to prior study withdrawal.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
percentage of participants
  GVHD-free Survival at 6 Months: number analyzed (Participants) | 53 | 63
  GVHD-free Survival at 6 Months | 45.3 [31.9 to 58.8] | 46.0 [33.7 to 58.3]
  GVHD-free Survival at 12 Months: number analyzed (Participants) | 53 | 63
  GVHD-free Survival at 12 Months | 50.9 [37.5 to 64.4] | 46.0 [33.7 to 58.3]
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with GVHD-free survival at 6 months post-randomization between the sirolimus and prednisone arms. These proportions were compared between treatment arms using a Z test of the difference of binomial proportions; Test type: Superiority; p = 0.936, Z test comparing binomial proportions — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: Sirolimus vs Prednisone; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.598, Z test comparing binomial proportions — Statistical significance was determined using a pre-specified threshold of 0.05

12. Secondary Outcome: Percentage of Participants With Serious Infections
Description: The cumulative incidence of serious infections (Grade 2 or 3 per BMT CTN MOP) is described, with death treated as a competing risk.
Time Frame: 6 and 12 Months Post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus | Prednisone
Number analyzed (Participants) | 58 | 64
percentage of participants
  Seirious Infections at 6 Months | 30.4 [18.9 to 42.7] | 43.8 [31.3 to 55.6]
  Seirious Infections at 12 Months | 39.6 [26.7 to 52.2] | 51.8 [38.8 to 63.4]
Statistical Analysis 1: Comparison: Sirolimus vs Prednisone; The null hypothesis is that there is no difference in the proportions of participants with serious infections between the sirolimus and prednisone arms during the 12 month period post-randomization, with death treated as a competing risk for serious infection. These proportions were compared between treatment arms using Gray's test; Test type: Superiority; p = 0.221, Gray's test — Statistical significance was determined using a pre-specified threshold of 0.05

ADVERSE EVENTS:
Time Frame: 1 Year Post-randomization
Arm/Group | Sirolimus | Prednisone
All-Cause Mortality (participants affected / at risk) | 12/58 | 17/64
Serious Adverse Events (participants affected / at risk) | 8/58 | 3/64
Other Adverse Events (participants affected / at risk) | 0/58 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=58) | Prednisone (N=64)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT02806947/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT02806947/SAP_001.pdf